CLINICAL TRIAL: NCT05981170
Title: To Evaluate the Impact of Home-based Adapted Physical Activity Programme for Patients With Brain Tumours and/or Metastatic Cancer Living in Rural Areas
Brief Title: Rurality Adapted Physical Activity Sport Health
Acronym: RAPASS
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Institut Cancerologie de l'Ouest (Other)
Responsible Party: Sponsor
Other Study IDs: ICO-2022-20
Record Dates: First submitted 2023-05-24; First posted 2023-08-08 (Actual); Last update posted 2023-08-08 (Actual); Status verified 2023-05

CONDITIONS: Brain Tumour; Metastatic Cancer
Keywords: Adapted physical activity; Rurality; Oncology; Physical fitness; Supportive care
MeSH Terms: conditions — Brain Neoplasms; Neoplasm Metastasis; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Adapted physical activity at home — The programme will take place over 6 months and will include :
  1 consultation with the oncologist who will first assess the need for Adapted Physical Activity and then prescribe the APA with a certificate of no physical contraindication
  1 consultation with the ICO's APA coach who will present the APA programme and assess the patient's physical capacity using the Short Physical Performance Battery (SPPB) test in order to adapt the programme to their needs.
  13 home-based APA sessions (ideally one session per week) with the EAPA from Departmental Committee for Sport for All in 49
  1 telephone call with the EAPA of the ICO to evaluate the programme 3 months after the last session.
  Patients will also be asked to complete questionnaires at the first session (S1), halfway through the sessions (S6) and at the last session (S13).
  These are FACIT-F 5Functional Assessment of Chronic Illness Therapy - Fatigue ; Ricci and L. Gagnon ; P-GIC (Patients' Global Impression of Change (PGIC) scale)

SUMMARY:
Physical activity (PA) has been an integral part of non-drug therapy since the early 2010s. This supportive care is likely to reduce fatigue and improve the quality of life of patients during and after the cancer treatment phase.

Physical activity also has a protective effect in terms of tertiary prevention by reducing the risk of recurrence of certain cancers (breast, colon, prostate) by around 40 to 50% and by reducing overall mortality.

Adapted physical activity (APA) is offered at the Institut de Cancérologie de l'Ouest (ICO) in Angers, but there are obstacles particularly linked to the geographical distance of the establishment where this activity is offered.

The RAPASS project is a prospective study which will be proposed to patients followed at the ICO, living in rural areas and far from Angers. Its main objective is to describe the fatigue and quality of life of patients before, during and after a 13-session home-based APA programme. The data collected will also be used to describe changes in physical condition and level, compliance with the programme, continuation of physical activity beyond the duration of the programme, and satisfaction.

DETAILED DESCRIPTION:
The oncologist first assesses the patient's need for APA. The patient is then seen by the ICO's APA coach (EAPA) who presents the APA programme. If the patient agrees to participate, the coach assesses the patient's physical capacity in order to adapt the programme to their needs.

The programme is then carried out with the departmental sports for all committee 49.

The frequency of practice will ideally be one session per week at the patient's home, supervised by a coach from Departmental Committee for Sport for All in 49. A total of 13 sessions will be carried out.

The sessions will aim to develop all the components of physical fitness (endurance, strength, balance, flexibility, coordination, etc.).

The patient receives a walking logbook to record the number of daily steps taken, an exercise booklet to work independently and a pedometer.

In the presence of the coach, the patients perform different exercises and complete different questionnaires.

The programme is evaluated by the ICO EAPA 3 months after the 13th and final session.

ELIGIBILITY:
Inclusion Criteria:

* Performans Status ≤ 2
* Patient living in a rural area
* Patient with a brain tumour and/or metastatic cancer
* Patient with a medical prescription for APA practice
* Patient with a certificate of no contraindication to physical activity

Exclusion Criteria:

* Persons deprived of their liberty, under court protection, under guardianship or under the authority of a guardian
* Patient unable to undergo the trial procedures for social or psychological reasons
* Patient who does not understand French

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients treated at the ICO Angers for a brain tumour and or metastatic cancer with medically measured APA needs.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2023-09 (Estimated); Primary Completion 2025-03 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Functional Assessment of Chronic Illness Therapy - Fatigue Scale (FACIT-F) | Through study completion, an average 6 months.
  To describe the fatigue (physical, functional, social, emotional components) of patients.
  The Score from FACIT-F range from 0 to 52. The higher the score, the lower is the fatigue.

SECONDARY OUTCOMES:
Short Physical Performance Battery test (SPPB) | Through studied intervention, an average 3 months.
  It is used to assess the physical performance of an individual. It is the result of the scores of three criteria: the balance test, the walking speed test and the chair lift test.
  The sum of the scores of all the tests gives an overall performance score:
  * SPPB 0-6: Poor performance
  * SPPB 7-9: Intermediate performance
  * SPPB 10-12: High performance
6 minute walk test | Through studied intervention, an average 3 months.
  This test measures the functional limitation by comparing the theoretical distance with the measured distance. The patient is asked to walk as far as possible within six minutes:
  * Excellent functional mobility ≥91% of the theoretical distance
  * Good functional mobility between 82% and 90% of the theoretical distance
  * Moderate functional limitation between 74% and 82% of the theoretical distance
  * Severe functional limitation ≤73% of the theoretical distance
Hand grip test | Through studied intervention, an average 3 months.
  This test measures muscular health of the hands and forearms.
Flexibility test | Through studied intervention, an average 3 months.
  The patient performs a standing trunk flexion with legs stretched. Depending on the area reached (hand touching the ground, kick, tibia, etc.), a score will be given on a scale of 1 to 5, which differs according to the patient's sex.
Balance test | Through studied intervention, an average 3 months.
  The patient is asked to stand on one leg for 1 minute with their eyes open. The best time is recorded and depending on the age and sex of the patient, his or her performance will be rated on a scale of 1 (very poor balance) to 4 (excellent balance).
Ricci et Gagnon questionnaire | Through study completion, an average 6 months.
  This questionnaire assesses the level of physical activity.
  A number of points ranging from 1 to 5 are assigned to each answer. The total sum of the points determines an overall score that classifies the patients into :
  * Score < 18 : inactive
  * 18 ≤ Score ≤ 35: active
  * Score > 35: very active
The Patient Global Impression scale (P-GIC) | At the end of the APA sessions, on average 3 months
  Evaluates the patient's satisfaction with the implementation of a home-based APA programme.
  The questionnaire includes a single question asking the patient what change home-based APA has had on their overall quality of life. The patient is given 7 options from which to choose the one that best corresponds to the perceived change: Very strongly positive, Strongly positive, Slightly positive, No change, Slightly negative, Strongly negative, Very strongly negative.

CONTACTS AND LOCATIONS:
Overall Officials: Loïc FAIVRE, Principal Investigator — Institut de Cancérologie de l'Ouest
Locations (1):
- Institut de Cancerologie de L'Ouest, Angers, France

IPD SHARING:
Plan to Share IPD: No